CLINICAL TRIAL: NCT06168565
Title: Hemodynamic Effects of Intermittent Pneumatic Compression for Sports: A Double-blinded Randomized Crossover Study
Brief Title: Hemodynamic Effects of Intermittent Pneumatic Compression for Sports
Acronym: IPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000001231
Record Dates: First submitted 2023-11-24; First posted 2023-12-13 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Sports Physical Therapy
Keywords: sports; recovery; intermittent pneumatic compression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Measures of end-diastolic peak velocity, systolic peak velocity, heart rate, and arterial diameter will be collected for two minutes, two minutes before, at the 8th minute after the start of the IPC administration, and two minutes after the conclusion of each IPC protocol. End-diastolic peak velocity and systolic peak velocity will be measured across different phases of the IPC cycle (all cuffs inflated, half of the cuffs inflated, and all cuffs deflated). Both the athletes and assessors will be unaware of which protocol is being carried out. All protocols will be performed with participants lying down in a supine position, on a stretcher. The moderate pressure protocol applies a pressure of 80mmHg and the high pressure protocol applies a pressure of 200mmHg.
  Interventions: Device: Intermittent pneumatic compression (AirRelax)
- Sequence 2 (Experimental): Measures of end-diastolic peak velocity, systolic peak velocity, heart rate, and arterial diameter will be collected for two minutes, two minutes before, at the 8th minute after the start of the IPC administration, and two minutes after the conclusion of each IPC protocol. End-diastolic peak velocity and systolic peak velocity will be measured across different phases of the IPC cycle (all cuffs inflated, half of the cuffs inflated, and all cuffs deflated). Both the athletes and assessors will be unaware of which protocol is being carried out. All protocols will be performed with participants lying down in a supine position, on a stretcher. The moderate pressure protocol applies a pressure of 80mmHg and the high pressure protocol applies a pressure of 200mmHg.
  Interventions: Device: Intermittent pneumatic compression (AirRelax)

INTERVENTIONS:
Device: Intermittent pneumatic compression (AirRelax) — Moderate pressure (around 80mmHg); high pressure (around 200mmHg), both applied on the lower-limbs
  Other Names: High pressure

SUMMARY:
The aim of this randomized crossover trial is to assess the hemodynamic effects caused by the use of 2 distinct intermittent pneumatic compression protocols on athletes.

The main questions it aims to answer are:

* Does intermittent pneumatic compression enhance athletes blood flow?
* If yes, what pressure is better to cause this enhancement?

ELIGIBILITY:
Inclusion Criteria:

* male gender
* healthy
* competing in soccer of track and field for at least two years
* not have performed any physical activity on the data collection day

Exclusion Criteria:

* more than one risk factor for thromboembolism (e.g., use of tobacco, varicose veins)
* injured athletes

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male gender
Enrollment: 23 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Arterial Diameter | 2 minutes before the IPC protocol, during (8th minute mark), and 2 minutes after the conclusion of the 15 minute protocol.
  Assessment of arterial diameter via automatic edge detection software (FMD Studio, Pisa, Italy) measuring the distance between the near and far wall of the intima
End-diastolic peak velocity | 2 minutes before the IPC protocol, during (8th minute mark - at different phases of the IPC cycle), and 2 minutes after the conclusion of the 15 minute protocol.
  End-diastolic peak velocity will be assessed in a supine position on the right common femoral artery using an ultrasound (Logiq e BT12; General Electric, Fairfield, CT, USA) with a 3 to 12 MHz multi-frequency linear phase array transducer.
Systolic peak velocity | 2 minutes before the IPC protocol, during (8th minute mark - at different phases of the IPC cycle), and 2 minutes after the conclusion of the 15 minute protocol.
  Systolic peak velocity will be assessed in a supine position on the right common femoral artery using an ultrasound (Logiq e BT12; General Electric, Fairfield, CT, USA) with a 3 to 12 MHz multi-frequency linear phase array transducer.

SECONDARY OUTCOMES:
Heart rate | 2 minutes before the IPC protocol, during (8th minute mark - at different phases of the IPC cycle), and 2 minutes after the conclusion of the 15 minute protocol.
  Assess any changes in heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Portugal